CLINICAL TRIAL: NCT06818552
Title: The Role of the Vascular Surgeon in Orthopedic Surgery of Musculoskeletal Tumors
Acronym: IOVA-mst
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IOVA-mst
Record Dates: First submitted 2024-11-28; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-10

CONDITIONS: Muscle Cancer
MeSH Terms: conditions — Muscle Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Very large musculoskeletal tumors frequently involve vascular structures. Literature data show that spinal surgery and orthopedic surgery are the specialist branches that most frequently require intraoperative vascular surgical assistance, with 33.8% and 26.4% of requests, respectively6.

In these cases, the surgical assistance of the vascular surgeon allows the safe removal of the mass, the possible repair of vessels damaged during cleavage and isolation of the mass, the ligation or complete reconstruction of the involved vascular segment and contributes to reducing intraoperative and postoperative complications7.

DETAILED DESCRIPTION:
Musculoskeletal tumors and spinal tumors represent a large and heterogeneous group of neoplasms. They are divided into primary soft tissue tumors (deriving from the neoplastic transformation of muscle, connective, vascular, lymphatic, nervous and adipose cells), primary bone tumors (deriving from the precursor cells of bone and cartilage cells) and spinal tumors. These neoplasms, depending on their location, can be either benign (chondroblastoma, chondromyxofibroma, enchondroma, fibrous dysplasia, benign giant cell tumor, non-ossifying fibroma, osteoblastoma, osteochondroma, osteoid osteoma, hemangioma, aneurysmal cyst, eosinophilic granuloma) or malignant (soft tissue sarcomas, osteosarcomas, chondrosarcomas, chondromas, Ewing's sarcoma, fibrosarcoma and undifferentiated pleomorphic sarcomas of the bone, myeloma/plasmacytoma, chordoma, meningioma, neurofibroma and schwannoma).

The initial presentation is frequently related to the mass effect that these tumors cause when they reach large dimensions. Equally often, particularly in the case of bone tumors, pain and pathological fractures represent the initial symptoms.

Both soft tissue and bone sarcomas are rare diseases with an incidence of 5 cases per 100,000 and 1 case per 100,000 inhabitants, respectively (data from AIRC - Italian Association for Cancer Research)1.

Due to their cellular heterogeneity, these tumors can be located in different areas of the human body, with a preference for the trunk and limbs; and they are often infiltrating in nature.

Their treatment is based, depending on the histotype and the degree of disease at the time of diagnosis, on surgical removal of the tumor, chemotherapy (CT), radiotherapy (RT) or a combination of these different methods.

The 5-year survival of these tumors varies, in addition to the histotype and degree, also on the experience of the center where the treatment takes place; and is estimated at around 70% for soft tissue sarcomas, 60% in localized forms of osteosarcoma and 80% in localized forms of chondrosarcoma2-4.

The radicality of the surgical treatment of these neoplasms is dictated in large part by obtaining wide resection margins that often involve surgical excisions extending beyond the structures directly involved by the tumor5.

Very extensive musculoskeletal tumors frequently involve vascular structures. Data from the literature show that spinal surgery and orthopedic surgery are the specialist branches that most frequently require intra-operative vascular surgical assistance, with 33.8% and 26.4% of requests, respectively6.

In these cases, the surgical assistance of the vascular surgeon allows the safe removal of the mass, the possible repair of the vessels damaged during the cleavage and isolation of the mass, the ligation or complete reconstruction of the involved vascular segment and contributes to reducing intra-operative and post-operative complications7.

The primary objective of the study is to evaluate the outcomes of the interventions for the removal of musculoskeletal tumors, in relation to the type of vascular surgical assistance provided.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with musculoskeletal tumor involving vascular structures requiring surgical removal
* Planned surgical treatment with intraoperative assistance of the vascular surgeon
* Obtaining informed consent
* Age 18 years

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with musculoskeletal tumor with involvement of vascular structures and indication for surgical treatment of removal of the mass that requires the presence of a vascular surgeon. This indication is supported by international guidelines and represents normal clinical practice in these patients.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of vascular issues during every procedure | From the first patient entrolled up to the 70th patient, up to 3 years
  Number of major and minor vascular complications are collected during every procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gargiulo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italia, Italy